CLINICAL TRIAL: NCT01182701
Title: Cognitive Behavioral Intervention in Diabetes Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Jillian Inouye/Principal Investigator, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 5R01NR007883 (NIH)
Record Dates: First submitted 2010-08-06; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Asian Pacific Islanders; Cognitive behavioral intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral intervention (Active Comparator)
  Interventions: Behavioral: Cognitive behavioral training
- Education support (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive behavioral training — The behavioral training group will be involved six group sessions focusing on cognitive behavioral training for stress and mood management, cognitive restructuring, empowerment, values clarification, problem solving and decision making via a manualized program
  Arms: Behavioral intervention

SUMMARY:
The proposed study is a two arm randomized controlled trial with longitudinal follow-up that compares cognitive behavioral interventions (ENHANCE) to a control group with attention. The experiment will consist of a repeated measure 2 X 3 design; Condition (Experiment vs. Control) by Time (Pre, Post, Follow Up).

ELIGIBILITY:
Inclusion Criteria:

* Asian/Pacific Islander Men and Women with type 2 diabetes; asymptomatic for hyperglycemia
* Both men and women will be included in the study if they have a diagnosis of type 2 diabetes made by a physician and meet classification and diagnostic criteria established by the American Diabetes Association (American Diabetes Association, 1997)
* Between 18 and 76 years
* Participation in diabetes education program of University Specialty Clinics

Exclusion Criteria:

* Crippling arthritis
* Joint replacements that limit movement
* Neuromuscular disease with paralysis
* Severe eye disease or visually impaired
* Chronic renal failure and/or End Stage Renal Disease requiring hemodialysis or peritoneal dialysis
* Transplant recipient
* Foot Amputation
* Congestive Heart Failure
* New York Heart Class III/IV
* Previous Cerebral Vascular Accident (stroke) with residual paralysis
* Malignancy
* Chronic hepatitis C
* HIV disease
* Individuals who contemplate changing residence within the period of study and becoming inaccessible to the study should be discouraged from the study

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2004-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Determine the effectiveness of a cognitive/behavioral intervention program in improving health outcomes of quality of life, general health, glycemic control, and depression. | Baseline
Determine the effectiveness of a cognitive/behavioral intervention program in improving health outcomes of quality of life, general health, glycemic control, and depression. | Post (6 weeks)
Determine the effectiveness of a cognitive/behavioral intervention program in improving health outcomes of quality of life, general health, glycemic control, and depression. | 6 months
Determine the effectiveness of a cognitive/behavioral intervention program in improving health outcomes of quality of life, general health, glycemic control, and depression. | 1 year

SECONDARY OUTCOMES:
Determine the effectiveness of a cognitive/behavioral intervention program in enhancing adherence to self-management strategies. | Baseline
Determine the effectiveness of a cognitive/behavioral intervention program in enhancing adherence to self-management strategies. | Post (6 weeks)
Determine the effectiveness of a cognitive/behavioral intervention program in enhancing adherence to self-management strategies. | 6 months
Determine the effectiveness of a cognitive/behavioral intervention program in enhancing adherence to self-management strategies. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Inouye, PhD, APRN, Principal Investigator — Universtiy of Hawaii
Locations (1):
- University of Hawaii School of Nursing & Dental Hygiene, Honolulu, Hawaii, United States